CLINICAL TRIAL: NCT01711736
Title: Immunogenicity and Safety Study of GSK Biologicals' Quadrivalent Influenza Vaccine (GSK2282512A) When Administered in Children
Brief Title: Study to Evaluate Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Influenza Vaccine GSK2282512A When Administered to Children 6 to 35 Months of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 116926; 2013-003155-38 (EudraCT Number)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Influenza
Keywords: Immunogenicity; Children; Safety; Seasonal influenza; Fluarix
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- GSK2282512A Group (Experimental): Subjects aged between 6 to 35 months inclusive received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of quadrivalent influenza GSK2282512A vaccine.
  Quadrivalent influenza GSK2282512A vaccine was administered intramuscularly in the left anterolateral thigh (subjects < 12 months of age) or the deltoid muscle (subjects ≥ 12 months of age).
  Interventions: Biological: Quadrivalent influenza GSK2282512A vaccine
- Fluarix Group (Active Comparator): Subjects aged between 6 to 35 months inclusive received 1 dose (primed subjects) at Day 0 and 2 doses (unprimed subjects) at Days 0 and 28 of Fluarix vaccine.
  Fluarix vaccine was administered intramuscularly in the left anterolateral thigh (subjects < 12 months of age) or the deltoid muscle (subjects ≥ 12 months of age).
  Interventions: Biological: Fluarix

INTERVENTIONS:
Biological: Quadrivalent influenza GSK2282512A vaccine — 1 or 2 doses administered intramuscularly (IM) in deltoid muscle or anterolateral thigh on Day 0 (primed subjects) and on Day 0 and Day 28 (unprimed subjects) respectively.
  Arms: GSK2282512A Group
Biological: Fluarix — 1 or 2 doses administered IM in deltoid muscle or anterolateral thigh, on Day 0 (primed subjects) and on Day 0 and Day 28 (unprimed subjects) respectively.
  Arms: Fluarix Group

SUMMARY:
The purpose of this study is to investigate the immunogenicity, reactogenicity and safety of the new influenza vaccine GSK2282512A (FLU-Q-QIV) and compare its activity to the marketed vaccine Fluarix® (TIV) in young children 6 to 35 months of age.

DETAILED DESCRIPTION:
The subjects will be randomized (1:1) in the 2 treatment groups to explore responses to vaccination in a sub-group analysis based on age (6 to 17 months, 18 to 35 months).

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* A male or female between, and including, 6 and 35 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Subjects in stable health as determined by the investigator's clinical examination and assessment of subject's medical history.
* Subjects are eligible regardless of history of administration of influenza vaccine in a previous season.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period. Routine registered childhood vaccinations are permitted.
* Child in care.
* Prior receipt of any seasonal or pandemic influenza vaccine within six months preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dosed.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of Guillain-Barré syndrome within six weeks of receipt of prior influenza vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Acute disease and/or fever at the time of enrolment.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 606 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2013-02-21 (Actual); Study Completion 2013-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Canada (6):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Santo Domingo, Distrito Nacional, Dominican Republic
- GSK Investigational Site, San Pedro Sula, Honduras

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bekkat-Berkani R, Ray R, Jain VK, Chandrasekaran V, Innis BL. Evidence update: GlaxoSmithKline's inactivated quadrivalent influenza vaccines. Expert Rev Vaccines. 2016;15(2):201-14. doi: 10.1586/14760584.2016.1113878. Epub 2015 Dec 5. PMID 26641539
- [Background] Langley JM, Wang L, Aggarwal N, Bueso A, Chandrasekaran V, Cousin L, Halperin SA, Li P, Liu A, McNeil S, Mendez LP, Rivera L, Innis BL, Jain VK. Immunogenicity and Reactogenicity of an Inactivated Quadrivalent Influenza Vaccine Administered Intramuscularly to Children 6 to 35 Months of Age in 2012-2013: A Randomized, Double-Blind, Controlled, Multicenter, Multicountry, Clinical Trial. J Pediatric Infect Dis Soc. 2015 Sep;4(3):242-51. doi: 10.1093/jpids/piu098. Epub 2014 Oct 20. PMID 26336604
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 116926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116926 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primed subjects: Received 2 doses of seasonal influenza vaccine separated by at least one month during the last season or had received at least 1 dose prior to last season. Unprimed subjects: Did not receive any seasonal influenza vaccine in the past or received only 1 dose for the first time in the last influenza season.
Pre-assignment Details: 5 subjects enrolled in the study were allocated subject numbers but the study vaccine dose was not administered.
Period: Overall Study
Arm/Group | GSK2282512A Group | Fluarix Group
Started | 299 | 302
Completed | 287 (Up to Day 180) | 294 (Up to Day 180)
Not Completed | 12 | 8
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Migrated/moved from study area | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2282512A Group | Fluarix Group | Total
Number analyzed (Participants) | 299 | 302 | 601
Age, Continuous [Mean (Standard Deviation); unit: Months] | 18.2 (8.17) | 18.1 (8.34) | 18.15 (8.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 146 | 301
  Male | 144 | 156 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Anti- Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains of Quadrivalent Influenza GSK2282512A Vaccine.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2), Flu B/Hubei-Wujiagang/158/09 (Yamagata) and Flu B/Bri/60/08 (Victoria). This outcome concerns solely subjects in the GSK2282512A Group.
Time Frame: At Day 28 for primed subjects and at Day 56 for unprimed subjects
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, in terms of antibody response measured by the Haemagglutination Inhibition assay, included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group
Number analyzed (Participants) | 284
subjects
  [H1N1, Day 28 = primed and Day 56 = unprimed] | 244
  [H3N2, Day 28 = primed and Day 56 = unprimed] | 205
  [Yamagata, Day 28 = primed and Day 56 = unprimed] | 224
  [Victoria, Day 28 = primed and Day 56 = unprimed] | 210

2. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain was defined as pain that prevented normal everyday activities. Grade 3 swelling was greater than 100 millimeters (mm) i.e. >100mm.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine administration documented.
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 291 | 297
subjects
  Any Pain | 95 | 91
  Grade 3 Pain | 7 | 3
  Any Redness | 6 | 6
  Grade 3 Redness | 0 | 0
  Any Swelling | 5 | 6
  Grade 3 Swelling | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms (Excluding Fever).
Description: Solicited general symptoms assessed were drowsiness, irritability/fussiness and loss of appetite. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 irritability/fussiness was defined as crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite was defined as not eating at all. Grade 3 drowsiness was defined as drowsiness that prevented normal activity.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 290 | 296
subjects
  Any Drowsiness | 93 | 88
  Grade 3 Drowsiness | 9 | 9
  Related Drowsiness | 79 | 80
  Any Irritability/fussiness | 118 | 123
  Grade 3 Irritability/fussiness | 15 | 14
  Related Irritability/fussiness | 104 | 106
  Any Loss of appetite | 99 | 100
  Grade 3 Loss of appetite | 16 | 14
  Related Loss of appetite | 84 | 83

4. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Fever
Description: Any fever was defined as any fever ≥38.0 degrees Celsius (°C) irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 fever was defined as fever ≥39.0 °C.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 290 | 296
subjects
  Any Fever | 61 | 60
  Grade 3 Fever | 23 | 13
  Related Fever | 49 | 48

5. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against Each of the Four Vaccine Influenza Strains
Description: HI antibody titres were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2), Flu B/Hubei-Wujiagang/158/09 (Yamagata) and Flu B/Bri/60/08 (Victoria)
Time Frame: At Day 0 (for all subjects) and 28 days after the last vaccine dose (at Day 28 for primed subjects and at Day 56 for unprimed subjects)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 284 | 287
Titers
  [H1N1, Day 0] | 9.6 [8.1 to 11.3] | 9.8 [8.3 to 11.6]
  [H1N1, Day 28 = primed and Day 56 = unprimed] | 157.1 [132.8 to 185.9] | 61.2 [49.2 to 76.2]
  [H3N2, Day 0] | 17.4 [14.1 to 21.5] | 13.8 [11.4 to 16.8]
  [H3N2, Day 28 = primed and Day 56 = unprimed] | 159.4 [129.4 to 196.3] | 103.0 [83.7 to 126.7]
  [Yamagata, Day 0] | 7.7 [6.9 to 8.7] | 7.2 [6.5 to 8.0]
  [Yamagata, Day 28 = primed and Day 56 = unprimed] | 114.2 [100.0 to 130.5] | 107.2 [92.2 to 124.6]
  [Victoria, Day 0] | 10.6 [9.1 to 12.4] | 9.3 [8.0 to 10.7]
  [Victoria, Day 28 = primed and Day 56 = unprimed] | 111.4 [91.9 to 135.2] | 15.6 [13.3 to 18.5]

6. Secondary Outcome: Number of Seroconverted Subjects for Anti- Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains of Fluarix Vaccine
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2), Flu B/Hubei-Wujiagang/158/09 (Yamagata) and Flu B/Bri/60/08 (Victoria). This outcome concerns solely subjects in the Fluarix Group.
Time Frame: At Day 28 for primed subjects and at Day 56 for unprimed subjects
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Fluarix Group
Number analyzed (Participants) | 287
subjects
  [H1N1, Day 28 = primed and Day 56 = unprimed] | 154
  [H3N2, Day 28 = primed and Day 56 = unprimed] | 160
  [Yamagata, Day 28 = primed and Day 56 = unprimed] | 222
  [Victoria, Day 28 = primed and Day 56 = unprimed] | 28

7. Secondary Outcome: Number of Subjects Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2), Flu B/Hubei-Wujiagang/158/09 (Yamagata) and Flu B/Bri/60/08 (Victoria)
Time Frame: At Day 0 (for all subjects) and Day 28 after last vaccine dose (Day 28 for primed subjects and Day 56 for unprimed subjects)
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 284 | 287
subjects
  [H1N1, Day 0] | 46 | 47
  [H1N1, Day 28 = primed and Day 56 = unprimed] | 254 | 169
  [H3N2, Day 0] | 93 | 74
  [H3N2, Day 28 = primed and Day 56 = unprimed] | 231 | 191
  [Yamagata, Day 0] | 26 | 24
  [Yamagata, Day 28 = primed and Day 56 = unprimed] | 242 | 229
  [Victoria, Day 0] | 56 | 45
  [Victoria, Day 28 = primed and Day 56 = unprimed] | 216 | 74

8. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Four Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum haemagglutination inhibition (HI) GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/CAL/7/09 (H1N1), Flu A/Victoria/361/11 (H3N2), Flu B/Hubei-Wujiagang/158/09 (Yamagata) and Flu B/Bri/60/08 (Victoria)
Time Frame: 28 days after the last vaccine dose (at Day 28 for primed subjects and at Day 56 for unprimed subjects)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 284 | 287
Fold increase
  [H1N1, Day 28 = primed and Day 56 = unprimed] | 16.4 [14.3 to 18.7] | 6.2 [5.3 to 7.3]
  [H3N2, Day 28 = primed and Day 56 = unprimed] | 9.1 [8.0 to 10.5] | 7.5 [6.4 to 8.7]
  [Yamagata, Day 28 = primed and Day 56 = unprimed] | 14.8 [12.8 to 17.1] | 14.8 [12.8 to 17.2]
  [Victoria, Day 28 = primed and Day 56 = unprimed] | 10.5 [9.2 to 11.9] | 1.7 [1.5 to 1.9]

9. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Fever
Description: Any fever was defined as any fever ≥38.0 °C irrespective of intensity and relationship to vaccination. Related was defined as symptoms considered by the investigator to have a causal relationship to vaccination. Grade 3 fever was defined as fever ≥39.0 °C.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 290 | 296
subjects
  Any Fever | 46 | 42
  Grade 3 Fever | 16 | 8
  Related Fever | 39 | 38

10. Secondary Outcome: Number of Subjects Reporting Any Medically Attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s).
Time Frame: During the entire study period (Day 0 to Day 180)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 299 | 302
subjects | 156 | 156

11. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) were defined as a subset of adverse events that included both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which might or might not have an autoimmune aetiology. Any pIMD was defined as at least one pIMD experienced by the study subject.
Time Frame: During the entire study period (Day 0 to Day 180)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 299 | 302
subjects
  Any pIMD(s) | 0 | 2
  Related pIMD(s) | 0 | 0

12. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: During the 28-day (Days 0-27) post-vaccination period.
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 299 | 302
subjects
  Any Unsolicited AEs | 142 | 165
  Grade 3 Unsolicited AEs | 9 | 5
  Related Unsolicited AEs | 17 | 13

13. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: as for outcome 2
Measure: Number; unit: subjects
Arm/Group | GSK2282512A Group | Fluarix Group
Number analyzed (Participants) | 299 | 302
subjects
  Any SAEs | 9 | 8
  Related SAEs | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 180; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events: During the 28-day (Days 0-27) post-vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | GSK2282512A Group | Fluarix Group
Serious Adverse Events (participants affected / at risk) | 9/299 | 8/302
Other Adverse Events (participants affected / at risk) | 200/299 | 211/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK2282512A Group (N=299) | Fluarix Group (N=302)
Bronchiolitis (Infections and infestations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 2
Amoebic dysentery (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Blastocystis infection (Infections and infestations) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Dengue fever (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Rotavirus infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK2282512A Group (N=299) | Fluarix Group (N=302)
Pain (General disorders) | 95 | 91
Drowsiness (General disorders) | 93/290 | 88/296
Irritability/fussiness (General disorders) | 118/290 | 123/296
Loss of appetite (General disorders) | 99/290 | 100/296
Fever (General disorders) | 61/290 | 60/296 — Assessed during the 7-day (Days 0-6) post-vaccination period
Fever (General disorders) | 46/290 | 42/296 — Assessed duringthe 4-day (Days 0-3) post-vaccination period
Nasopharyngitis (Infections and infestations) | 78 | 90
Diarrhoea (Gastrointestinal disorders) | 38 | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.